CLINICAL TRIAL: NCT07183150
Title: A Single Center, Prospective Study on the Possible Range of No.4sb Lymph Node Dissection of Locally Advanced Distal Gastric Cancer
Brief Title: The Possible Range of No.4sb Lymph Node Dissection of Locally Advanced Distal Gastric Cancer
Acronym: Range of 4sb
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E20250853
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Gastric Cancer (GC); No.4sb
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The reasonable range of No.4sb lymph node dissection: The No.4sb lymph node divided into the lymph nodes on the root of left gastric omentum vessels (No.4sb-R) and the lymph nodes on the greater curvature side (No.4sb-C). Observation of lymph node metastasis rates in two groups.

SUMMARY:
The main purpose of this study is to evaluate the reasonable range of No.4sb lymph node dissection of locally advanced distal gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 and ≤ 75 years of age; Preoperative gastric cancer patients with pathologically confirmed; Had been treated with Radical resection (D2, R0) of gastric cancer (Lymph node≥16); Willing and able to comply with the program during the study period; Physical condition and organ function allows to tolerable abdominal surgery; Written informed consent provided; Under radical laparoscopic distal subtotal gastrectomy With more than a 6-month life expectancy; No other serious concomitant diseases; Sufficient organ functions; No previous history of chemotherapy or radiotherapy; Clinical stage: T2-4aNxM0; Karnofsky performance status (KPS)>60; Eastern Cooperative Oncology Group Performance Status (ECOG): 0-1.

Exclusion Criteria:

Pregnancy or breast feeding; Patients with Serious liver disease (such as cirrhosis, etc.), kidney disease, respiratory disease or uncontrolled diabetes, hypertension and other chronic systemic diseases, heart disease with Clinical symptoms, such as congestive heart failure, coronary heart disease symptoms, drug is difficult to control arrhythmia, hypertension, or six months had a myocardial infarction attack, or cardiac insufficiency; Organ transplantation patients need immunosuppressive therapy; Severe recurrent infections were not controlled or with other serious concomitant diseases; Patients got other primary malignant tumors (except curable skin basal cell carcinoma and cervical cancer in situ) except gastric cancer within 5 years; Psychiatric disease which require treatment; Have the history of organ transplantation; Within 6 months before study starts and in the process of this study, patients participate in other clinical researches.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 patients with advanced gastric cancer，underwent radical laparoscopic distal gastrectomy. Observation of lymph node metastasis in different No.4sb subgroups.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-08-17 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The lymph node metastasis rates in No.4sb-R, No.4sb-C and No.4d groups. | 400 cases enrolled within 3 years
  Observation of lymph node metastasis in No.4sb-R, No.4sb-C and No.4d groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China